CLINICAL TRIAL: NCT00386919
Title: A Phase II Study of Hypofractionated Radiation With CyberKnife Stereotactic Radiosurgery Boost for High Grade Gliomas in Elderly Patients With Good Performance Status
Brief Title: Short Course of Radiation for Gliomas in Elderly Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Anand Mahadevan, Radiation Oncologist, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006P-000110/3
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: High Grade Gliomas
MeSH Terms: interventions — Radiosurgery

INTERVENTIONS:
Procedure: CyberKnife

SUMMARY:
Patients with high grade brain tumors will be treated to test shortened course of radiation therapy with the use of precise, focused radiation with cyberknife.

DETAILED DESCRIPTION:
Screening Procedures: Screening procedures are tests and procedures that will be done to determine if you are eligible to take part in the research study. For this research study, the screening procedures include: Medical history, physical examination including neurological and performance status, assessment of preoperative and postoperative scans, operative reports and pathology reports. All of these have already been performed or will be performed as standard of care for your condition even if you are not taking part in this study.

Research Procedures: If you qualify to take part in this research study, you will undergo these research procedures: The pre- and post operative MRI (Magnetic Resonance Imaging) scans before and after your operation, the operative procedure (including sampling known as biopsy or removal of as much as tumor as possible) and the procedures to facilitate radiation therapy planning (making a mask in the treatment position to keep you comfortably still and CAT scan in the treatment position). These are all part of standard procedures in the treatment of your tumor, whether you are in this study or not.

One of the primary reasons to deliver radiation in multiple small doses conventionally (30-33 treatments over 6-61/2 weeks) is to minimize damage to the surrounding normal brain. The Cyberknife technology allows precise delivery of radiation to your tumor while minimizing radiation to the surrounding brain. This allows the possibility of delivering higher doses of radiation to the tumor thereby shortening the overall treatment time (18 treatments in 31/2 weeks). This is what is being studied in this study.

The Cyberknife treatment will be longer in duration lasting about 30-60 minutes rather than 5-10 minutes with each conventional radiation treatment. During this time you will be asked to lie as comfortably still as you can. The technology however permits the radiation beam to adjust precisely to any small movements you may make to maintain the accuracy.

Along with radiation, you will get chemotherapy called Temozolomide, in the form of pills. This is also standard treatment whether or not you are in this study. You will be asked to take these pills every day during the course of radiation and for 5 days each month thereafter for a year. However during radiation you will be receiving Temozolomide, which is used to possibly make the radiation more effective, only for 4 weeks as opposed to 6 weeks of conventional radiation. As part of usual care with this chemotherapy you may receive supportive medication to prevent and treat nausea, vomiting, low blood counts or infection.

Monitoring/Follow-Up Procedures. Procedures performed to evaluate the effectiveness and safety of the experimental procedures are called "monitoring" or "follow-up" procedures. For this research study, the monitoring/follow-up procedures include: Clinical assessment including neurological and performance status assessments and blood tests for your chemotherapy will be performed every month for the first year and every three months thereafter. MRI scans one month after completion of radiation therapy and every 2 months thereafter. All these procedures are performed routinely in the management of your tumor

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed High Grade Glioma (oligo-, astro- or mixed gliomas).
* >65 years of age
* KPS>70
* No contraindication for Radiation or Chemotherapy
* Histopathologically confirmed newly diagnosed glioblastoma multiforme or Anaplastic Glioma (WHO Grade III) by surgical excision or biopsy.
* Patient must have recovered from the effects of surgery, post-operative infection, or other complications.
* Therapy should start within 5 weeks of surgery
* Must have an estimated survival of > 8 weeks.
* KPS > 70.
* Age > 65 years.
* Must have a pre- and post operative contrast enhanced MRI scans
* Laboratory values within the following limits: ANC (absolute neutrophil count) >/= 1.5x 109/l, Platelets >/= 100x 10 9 /L, Hemoglobin >/= 9g/dl, Serum Creatinine >/= 1.5mg/dl., Serum total Bilirubin </= 1.5 x upper limit of normal (ULN), SGOT/SGPT </= 2.5x ULN, Albumin >/= 3g/dl.
* If the patient receiving an enzyme inducing antiepileptic drug will be switched to an NEIAED (Non Enzyme Inducing Anti Epileptic Drug).

Exclusion Criteria:

* Histology grade less than Anaplastic Glioma ( WHO Grade III).
* Recurrent malignant glioma.
* Tumor involving the Brain stem.
* Any detected tumor foci beyond the cranial vault.
* Major medical or psychiatric illness, which in the investigator's opinion will prevent administration or completion of the protocol therapy.
* Prior malignancies, except for non-melanomatous skin cancers, or carcinoma in situ of uterus, cervix or bladder, unless disease free for > 5 years.
* Prior radiation to the head or neck (except for T1 glottic cancer) resulting in overlap of radiation fields.
* Prior chemotherapy for the current disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability of short duration involved field radiation followed by CyberKnife Radiosurgery Boost | 1 month

SECONDARY OUTCOMES:
Assessment of local control rate, progression free survival, overall survival, quality of life and toxicity and steroid dependence in this population with this regime | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anand Mahadevan, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States